CLINICAL TRIAL: NCT01022242
Title: A Prospective Double-blind, Randomised Concept Study of PXL01 Versus Placebo in Flexor Tendon Surgery
Brief Title: Study of PXL01 Versus Placebo to Inhibit Adhesion Formation After Flexor Tendon Surgery
Acronym: PHSU02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pergamum AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PHSU02
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Results first posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-04

CONDITIONS: Surgical Adhesions
Keywords: Surgical Adhesions; Post-surgical adhesions; Flexor tendon
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo is administered locally between the flexor tendon and the tendon sheath and around the tendon sheath at a volume of 0.5 ml. Administration of the product is carried out after repair of the flexor tendon but before closure of the surgical wound.
  Interventions: Drug: Placebo
- PXL01 (Experimental): PXL01 is administered locally between the flexor tendon and the tendon sheath and around the tendon sheath at a volume of 0.5 ml. Administration of the product is carried out after repair of the flexor tendon but before closure of the surgical wound.
  Interventions: Drug: PXL01

INTERVENTIONS:
Drug: PXL01 — PXL01 is a synthetic peptide sequentially derived from human lactoferrin. PXL01 is formulated in a viscous solution of sodium hyaluronate. The drug product is administered locally between the flexor tendon and the tendon sheath and around the tendon sheath at a volume of 0.5 ml. Administration of the product is carried out after repair of the flexor tendon but before closure of the surgical wound.
  Arms: PXL01
Drug: Placebo — Placebo is a physiological sodium chloride solution, which is clear and colourless.
  Arms: Placebo

SUMMARY:
The objectives of the study are to assess efficacy, safety, and handling of PXL01 in patients with flexor tendon injury in zone I or II.

DETAILED DESCRIPTION:
This is a multi-centre, randomized, double blind, parallel study design in patient admitted for flexor tendon repair in zone II.

The patients will undergo 9 visits within the time frame of the study. Patients will be randomized to receive treatment with PXL01 or standard care.

Primary objective is to assess total active motion based on PIP and DIP joints (TAM2) at 12-week visit. Secondary objectives are to assess TAM2 at all time points except for 12 weeks, TAM based on MCP, PIP, and DIP joints (TAM3) at all time points, Total Active Motion in DIP joint (DIPAM), tip-to-crease, grip strength and Total Passive Motion (TPM2 and TPM3).

Before any study-related assessment takes place, patients are given verbal and written information about the study and informed consent is achieved from the patient and/or legal guardian. The study should be carried out in accordance with the Clinical Study Protocol (CSP), ICH guidelines for Good Clinical Practise (GCP), and applicable regulatory requirements.

ELIGIBILITY:
Inclusion criteria:

1. Complete division of flexor digitorium profundus tendon (FDP) in zone I or II, with or without division of flexor digitorium superficialis (FDS) and possible to rejoin with tendon suture
2. Open flexor tendon injury sutured within 14 days after trauma
3. 12-75 years of age
4. Signed informed consent prior to any study related procedures

Exclusion criteria

1. Treatment with any investigational product within 4 weeks of study entry
2. Patients previously included in the study
3. Thumbs with complete or partial division of flexor pollicis longus (FPL)
4. Concomitant fracture(s) requiring immobilisation
5. Injuries with associated soft tissue loss
6. Severe crush injury
7. Palmar plate injury requiring immobilisation
8. Devascularisation/requirement of vascular repair
9. Joint injuries
10. Bilateral injuries
11. Previous flexor tendon surgery in the digit, which is to be treated with IMP
12. Reduced motion in the digit, which is to be treated with IMP, or the corresponding digit prior to the injury
13. Compliance with mobilisation protocol not expected
14. Alcohol or drug abuse
15. Severe intercurrent illness, which in the opinion of the Investigator, may put the patient at risk when participating in the study, or affect the patient's ability to take part in the study
16. Pregnant or lactating females
17. Fertile women who do not accept the consistent and correct use of highly effective methods of birth control defined as implants, injectables, combined oral contraceptives, intra-uterine device (IUD)s, sexual abstinence or vasectomised partner during the first two weeks post-surgery. A condom alone is not considered an acceptable method for birth control, not even together with spermicide.
18. Known allergy to any component of the study product or placebo
19. Patients suffering from:

    * Diabetes Mellitus patients where significant diabetic complications may delay healing according to the investigator's judgement
    * Rheumatoid arthritis
20. Or patients treated with:

    * Systemic steroids within one month
    * Immunosuppressive drugs within three months
    * Daily use of NSAIDs within one week or occasional use within 8 hours

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2009-12; Primary Completion 2012-05 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Wiig, MD, PhD, Principal Investigator — Dept. of Hand Surgery Uppsala University Hospital
Locations (15):
- Denmark (2):
  - Dept. of Hand Surgery, Aalborg Hospital, Aalborg
  - Dept. of Hand Surgery, Odense University Hospital, Odense
- Germany (9):
  - Klinik für Handchirurgie der Herz- und Gefäß-Klinik GmbH, Bad Neustadt an der Saale
  - Katholisches Klinikum Duisburg, St. Barbara Hospital, Klinik für Plastische Chirurgie und Handchirurgie, Duisburg
  - St.Josef Hospital Essen- Kupferdreh, Abteilung für Handchirurgie, Essen
  - Klinik für Plastische, Hand- und Wiederherstellungschirurgie, Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum des Saarlandes, Klinik für Unfall-, Hand - und Wiederherstellungschirugie, Homburg
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Sektion für Plastische Chirurgie, Handchirurgie und Intensiveinheit für Schwerbrandverletzte, Lübeck
  - Ludwig-Maximilians Universität München, Klinik und Poliklinik für Plastische Chirurgie und Handchirurgie, Campus Innenstadt, Munich
  - Ludwig-Maximilians Universität München, Klinik und Poliklinik für Plastische Chirurgie und Handchirurgie, Campus Großhadern, Munich
  - Klinik für Handchirurgie, Mikrochirurgie und Rekonstruktive Brustchirurgie Vinzenz von Paul Kliniken GmbH, Stuttgart
- Sweden (4):
  - Dept. of Hand Surgery Sahlgrenska University Hospital, Gothenburg
  - Dept. of Hand Surgery Malmö University Hospital, Malmo
  - Dept. of Hand Surgery, Stockholm South General Hospital, Stockholm
  - Dept. of Hand Surgery Uppsala University Hospital, entrance 70, Uppsala

REFERENCES:
- [Derived] Wiig ME, Dahlin LB, Friden J, Hagberg L, Larsen SE, Wiklund K, Mahlapuu M. PXL01 in sodium hyaluronate for improvement of hand recovery after flexor tendon repair surgery: randomized controlled trial. PLoS One. 2014 Oct 23;9(10):e110735. doi: 10.1371/journal.pone.0110735. eCollection 2014. PMID 25340801

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | PXL01
Started | 70 (71 pat rand to placebo. 1 got incorrect mix of placebo. 70 patients treated with the correct mix.) | 65 (67 pat rand to PXL01. 2 got incorrect mix of PXL01. 65 patients treated with the correct PXL01 mix.)
Completed | 49 | 46
Not Completed | 21 | 19

BASELINE CHARACTERISTICS:
Population: 3 patients were treated with an incorrect mixture of IMP and were analyzed separately.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PXL01 | Total
Number analyzed (Participants) | 70 | 65 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 4 | 6
  Between 18 and 65 years | 66 | 60 | 126
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 51 | 48 | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 64 | 62 | 126
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: TAM2
Description: The primary variable is TAM2: The sum of Total Active Motion at the proximal interphalangeal (PIP) and distal interphalangeal (DIP) joints of the affected digit at actively made fist minus the extensor lag at these joints.
Time Frame: At 12 weeks after surgery
Population: FAS population
Measure: Median (Full Range); unit: Degrees
Arm/Group | Placebo | PXL01
Number analyzed (Participants) | 51 | 50
Degrees | 108 [36 to 175] | 121 [29 to 182]
Statistical Analysis 1: Comparison: Placebo vs PXL01; Test type: Superiority or Other; p = 0.8861, ANCOVA

ADVERSE EVENTS:
Arm/Group | Placebo | PXL01
Serious Adverse Events (participants affected / at risk) | 9/70 | 10/65
Other Adverse Events (participants affected / at risk) | 22/70 | 22/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=70) | PXL01 (N=65)
Tendon rupture (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
allergic urticaria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
syncope (Nervous system disorders) | 1 (1) | 0 (0)
adhesion (resulting in tenolysis) (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
accidental death (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
myeloproliferative disorder (Immune system disorders) | 0 (0) | 1 (1)
stroke (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=70) | PXL01 (N=65)
Oedema peripheral (General disorders) | 4 (5) | 5 (5)
Nasopharyngitis (Infections and infestations) | 8 (8) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Localised Infections (Infections and infestations) | 2 (2) | 4 (4)

LIMITATIONS AND CAVEATS:
High drop out rate leading to a low number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less